CLINICAL TRIAL: NCT03770663
Title: Cyclophosphamide and Azathioprine vs Tacrolimus in Antisynthetase Syndrome-related Interstitial Lung Disease : Multicentric Randomized Phase III Trial
Brief Title: Cyclophosphamide and Azathioprine vs Tacrolimus in Antisynthetase Syndrome-related Interstitial Lung Disease
Acronym: CATR-PAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140217; 2016-002921-12 (EudraCT Number)
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Antisynthetase Syndrome (ASS); Interstitial Lung Disease
MeSH Terms: conditions — Antisynthetase syndrome; Lung Diseases, Interstitial | interventions — Cyclophosphamide; Azathioprine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- European strategy (Experimental): 3 IV pulses of Methylprednisolone (7.5 mg/kg/day followed by tapering doses of oral Prednisone, started at 1 mg/kg/day from D4 to M12
  In association with:
  6 IV pulses of Cyclophosphamide (1000mg) followed from M5 to M12 by oral Azathioprine (2mg/kg/day), with a maximum of 150mg/day
  Interventions: Drug: Cyclophosphamide and azathioprine
- American strategy (Experimental): 3 IV pulses of Methylprednisolone (7.5 mg/kg/day followed by tapering doses of oral Prednisone, started at 1 mg/kg/day from D4 to M12
  In association with:
  Tacrolimus given orally from M0 to M12 (started at the initial dose of 2x2mg/day). Tacrolimus doses are regularly adapted to its serum concentration to reach 5-15ng/mL.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclophosphamide and azathioprine — European strategy 6 IV pulses of Cyclophosphamide (1000mg) followed from M5 to M12 by oral Azathioprine (2mg/kg/day), with a maximum of 150mg/day
  Arms: European strategy
Drug: Tacrolimus — American strategy Tacrolimus given orally from M0 to M12 (started at the initial dose of 2x2mg/day). Tacrolimus doses are regularly adapted to its serum concentration to reach 5-15ng/mL.
  Arms: American strategy

SUMMARY:
"Antisynthetase syndrome (ASS) is one of the most severe inflammatory myopathy (IM), due to pulmonary involvement (interstitial lung disease, ILD). Until now, the most commonly used immunosuppresive therapy in Europe is Cyclophosphamide followed by different immunosuppressive drugs as maintenance therapy, including Azathioprine (and so called " European Strategy "). In the USA however, the first-line immunosuppressive treatment is Tacrolimus (so called " American Strategy "). None of these two different strategies has ever been studied prospectively, and there is no clear comparison of short and long-term treatment efficacy and tolerance. Thus, there are yet no evidences helping the clinicians in the therapeutic management of patients with ASS-related ILD.

The aim of this study is therefore to compare both strategies as first line treatments or in relapsing patients : CATR.PAT study is a 52 weeks, randomized, comparative, controlled, open-labeled, phase III, therapeutic clinical trial, comparing two treatment strategies."

DETAILED DESCRIPTION:
"During the study period, according to randomization into two groups (n=38 patients, respectively), patients will receive either:

- Group 1 & 2 : 3 IV pulses of Methylprednisolone (7.5 mg/kg/day followed by tapering doses of oral Prednisone, started at 1 mg/kg/day from D4 to M12

In association with :

* Group 1 : European Standard of care :

  6 IV pulses of Cyclophosphamide (1000 mg) followed from M5 to M12 by oral Azathioprine (2 mg/kg/day), with a maximum of 150 mg/d)
* Group 2 : American Strategy Tacrolimus is given orally from M0 to M12 (started at the initial dose of 2x2mg/d). Tacrolimus doses are regularly adapted to its serum concentration to reach 5-15 ng/ml."

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Signed informed consent
3. Affiliation to the Social security system
4. Diagnosis of ASS: positive test for any of the 5 anti-tRNA synthetase antibodies routinely tested (ELISA, Luminex or Linear-dot), including anti-Jo-1, anti-PL7, anti-PL12, anti-EJ and anti-OJ.
5. Diagnosis of ILD-related ASS: interstitial lung disease on HRCT.
6. Moderate to severe ILD on PFT : FVC < 80% and or cDLCO < 70%
7. beta-HCG test negative or negative uterine echography (for women of child bearing potential)
8. Women of childbearing potential must have an oral contraception (macroprogestatifs) during all the duration of study treatment and 12 months after the last dose of study treatment
9. Males who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of study treatment and 6 months after the last dose of study treatment

Exclusion Criteria:

1. Pregnancy and/or breast feeding
2. Others contraindications to the treatments, including hypersensitivity to the drug (including excipient and active compounds), medical contraception contraindications, severe renal failure, severe hepatic insufficiency and severe psychiatric disorders. Specific contraindications are listed for each experimental medication in Table 6 (according to updated Summary of product characteristics, see Appendix 8)
3. Fever or active bacterial infection (ie. septicemia, pneumopathy, pyelonephritis, acute prostatitis …), or parasitic infection (ie. Anguillulosis …),or fungal infection (ie. Invasive pulmonary aspergillosis …), or viral infection (HIV seropositivity, Active Tuberculosis, active B/C viral hepatitis, CMV, active EBV…)
4. Active neoplasm
5. Previous inefficacy of Cyclophosphamide, Azathioprine or Tacrolimus, not related to adhesion problems.
6. Previous use of 3 daily IV steroids < 3 months before patient's enrollment.
7. ASS-related ILD worsening or relapse under Prednisone > 0.5 mg/kg/day
8. Previous use of Cyclophosphamide, Azathioprine or Tacrolimus in the last 6 months.
9. Severe ASS requiring ICU (respiratory disease, myocarditis), plasma exchange or IV-Ig.
10. Positivity of auto-antibodies associated to Systemic Sclerosis (anti-Telomerase, anti-Centromères, anti-Polymerase III).
11. Patients with QTc > 450 msec
12. Patients with history of long QT syndrome (including familial) or ventricular arrhythmias
13. Concomitant use of drugs prolonging QT / QTc (list of treatments in annex)
14. Hypokalemia
15. Patients with pulmonary hypertension detected on echocardiography during the screening/selection visit (systolic pulmonary artery pressure (PAP) was 37-50 mmHg, and/or tricuspid regurgitation velocity 2.8-3.4 ms-1) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From baseline to 12 months
  Compare the efficacy of Cyclophosphamide and Azathioprine vs Tacrolimus in patients with ASS related-ILD Time from the initiation of treatment to the first event related to ASS related-ILD (progression free survival)

SECONDARY OUTCOMES:
Variation of the six minute walk tests | at baseline, 3 months, 6 months, 9 months and 12 months
  Compare Global variation of the M0 and M12-six minute walk tests (distance in meter, differential of saturation in %)
Forced Vital Capacity (FVC) | at baseline, 3 months, 6 months, 9 months and 12 months
  Compare Global variation of M0 and M12-FVC (both absolute and %)
Diffusing Lung Carbon Monoxyde Capacity (cDLCO) | at baseline, 3 months, 6 months, 9 months and 12 months
  Compare Global variation of M0 and M12 cDLCO (both absolute and %)
Rate of pulmonary improvement | at baseline, 3 months, 6 months, 9 months and 12 months
  Lung improvement is defined (in the absence of any other pulmonary disease) by 3A. Improvement of at least 20% of the dyspnea visual scale score (1-10) 3B. and/or improvement of pulmonary function tests: increase of the baseline FVC by 10% (% patient predicted value or absolute value) or of the baseline cDLCO by 15% (% patient predicted value or absolute).
  3C. and/or improvement of ILD on HRCT-scan (-5% involvement of the lung parenchyma evaluated by the extension score and -10% of the coarseness score of fibrosis): see Appendix 3' 3D. and/or improvement of PaO2 > 10 mmHg (FiO2=21%), without hyperventilation at any test
Time to extra-pulmonary improvement | at each visits
  Evaluated as follow :
  4A. improvement of the muscle involvement assessed by muscle manual testing (MMT/150, see Appendix 5) at each visit, is defined by an increased score > 20% 4B. biological improvement of the muscle involvement, assessed by creatine kinase levels performed at every visit, is defined by a decreased of baseline creatin kinase > 50% (IU/ml) 4C. improvement of the joint involvement, assessed by the ACR score at every visit is defined by a decrease > 20% of baseline number of swelling and painful joints.
Rate of extra-pulmonary improvement | at baseline and 12 months
  Extra-pulmonary improvement (muscle and joint involvements) is evaluated as follows :
  5A. improvement of the muscle involvement, assessed by MMT/150 muscle testing at baseline and M12, is defined by an increased score > 20% 5B. improvement of the joint involvement, assessed by the ACR score at each visit is define by a decrease > 20% of baseline number of swelling and painful joints.
Treatments tolerance | At every visit
  6A. any serious adverse event attributable to any experimental medication, which requires hospitalization, is recorded at any time 6B. side effects are declared by the patients, recorded and reported by the investigators at every visit 6C. the number of patients switching of experimental treatment is recorded 6D. the cumulative dose (mg/kg) of steroids will be compared at the end of the study
Treatment Efficacy | at every visit
  6A. any serious adverse event attributable to any experimental medication, which requires hospitalization, is recorded at any time 6B. side effects are declared by the patients, recorded and reported by the investigators at every visit 6C. the number of patients switching of experimental treatment is recorded 6D. the cumulative dose (mg/kg) of steroids will be compared at the end of the study
Quality of Life with SF-36 scale | Baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire Pitié Salpêtrière, Paris, France